CLINICAL TRIAL: NCT04260646
Title: Enuresis Alarm for Treatment of Urinary Incontinence in Children With Combined Daytime Incontinence and Enuresis
Brief Title: Alarm Treatment for Combined Enuresis and Daytime Urinary Incontinence in Children
Acronym: ABDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Regional Hospital West Jutland (Other); Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Søren Hagstrøm, MD PhD, Consultant, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20170005
Record Dates: First submitted 2019-07-18; First posted 2020-02-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Incontinence, Urinary; Enuresis, Nocturnal; Enuresis
MeSH Terms: conditions — Urinary Incontinence; Nocturnal Enuresis; Enuresis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Urotherapy without enuresis alarm (Active Comparator): Standard urotherapy inclunding normalized fluid intake and times voidings. The timed voiding regime of every 2 hours will be assisted by a timer Watch.
  Interventions: Device: Timer watch (Rodger)
- Standard Urotherapy with enuresis alarm (Experimental): Standard urotherapy inclunding normalized fluid intake and times voidings. The timed voiding regime of every 2 hours will be assisted by a timer Watch. In addition an enuresis alarm will be provided and worn by the participants during the night.
  Interventions: Device: Enuresis Alarm Rodger and Timer watch (Rodger); Device: Timer watch (Rodger)

INTERVENTIONS:
Device: Enuresis Alarm Rodger and Timer watch (Rodger) — Nocturnal enuresis fluid sensitive alarm and Timer watch (Rodger) vibrating or sounding alarm for remembering timed voiding intervals
  Arms: Standard Urotherapy with enuresis alarm
Device: Timer watch (Rodger) — Timer watch (Rodger) vibrating or sounding alarm for remembering timed voiding intervals

SUMMARY:
The aim is to examine whether alarm therapy in addition to urotherapy can have a beneficial effect in treating urinary incontinence children with combined daytime incontinence and enuresis. The study will include children who suffers for combined daytime incontinence and enuresis and referred to one of the pediatric departments were offed to participate. Participants are randomized to 8 weeks treatment with either enuresis alarm and timer watch assist urotherapy or solely timer watch assisted urotherapy.

DETAILED DESCRIPTION:
Urinary incontinence are common disorders of school age children. Approximately 3.8 - 16.9 % of first grade children suffer from daytime incontinence (DUI) depending on the definitions. Half of the children with DUI suffers for enuresis (NE) too. The background for combined DUI and enuresis is in most children functional overactive bladder (OAB).

At present DUI is treated first with urotherapi, if insufficient bladder modulating drugs are added. When daytime continence is achieved, the enuresis is handled using (in cases of small bladder capacity) an enuresis alarm.

Whether daytime continence is a prerequisite for treating NE or whether enuresis alarm may positively influence DUI treatment has not been studies in a RCT previously.

The aim of this study is to examine whether alarm therapy in addition to urotherapy can have a beneficial effect in treating children with combined daytime incontinence and enuresis. Thus the hypothesis are:

1. That the enuresis alarm therapy is beneficial in DUI treatment.
2. That it is possible to treat enuresis before daytime continence has been achieved

Methods: The study is a randomized controlled trial. The participants will be approx. 90 children that suffers from combined enuresis and daytime urinary incontinence. The participants will be equally randomized to 8 week of timer watch assisted urotherapy 1) with or 2) without addition of enuresis alarm treatment. The study includes 3 outpatient visits and 2 phone contacts.

The participants will complete bladder diaries as well as drypie and nocturnal urine production registrations. Also registrations on number and time of enuresis will be recorded for the alarm group children. All children will be provided a timer watch.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-14 years
* Completed "Tørfisk" (Danish version of the Bower "Dry pie" Incontinence diary 1) and bladder diary (containing frequency and volume of voiding, fluid intake through 48 hours as well as 7 days night registering of nocturnal urine production (NUP) and wet nights.)
* A minimum of 2 wet days per week
* A minimum of 2 wet nights per week.
* Average NUP (aNUP) on wet nights of less than 130 % of expected bladder capacity (EBC=30*(age+1))
* Obtained oral and written informed consent from the participant and both custody holders.

Exclusion Criteria:

* Known renal- or urinary tracts anomalies that affects the incontinence
* Ongoing urinary tracts infection (UTI)
* Ongoing obstipation defined by ROM IV criteria
* Glycosuria or proteinuria
* Previously received treatment with anticholinergics
* Previously received treatment with enuresis alarm
* Sign on neurological or structural cause of the incontinence
* Reduced compliance for alarm treatment defined as use of the alarm less than 80 % of the nights of the treatment period.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Daytime incontinence-score | Score will be calculated pre intervention, at week 2, 4, 6, and 8 of intervention
  Incontinence-score calculated from Drypie scale between 0-21
Change in Relative number of wet nights | Will be calculated from registrations at baseline and week 8 of intervention
  Number of wet nights pr week

SECONDARY OUTCOMES:
Change in MVV (maximal voided volume) | Will be calculated from 48h registrations at baseline and at week 8 of intervention
  maximal voided volume from bladder diary in ml
Change in Daytime urinary incontinence episodes (DUI episodes) | Will be calculated from 48h registrations at baseline and at week 8 of intervention
  Daytime urinary incontinence episodes by bladder diary (episodes per day)

OTHER OUTCOMES:
Change in fluid intake | Change in Fluid intake from 48h registrations at baseline and week 8 of intervention
  fluid intake from bladder diary (ml fluid per day)
Change in enuresis time | Change in timepoint of enuresis from week1 to week8
  time of enuresis during night (timepoint)
Change in number of enuresis episodes | Change in number of weekly enuresis measured one week at Baseline (before intervention) and week 8 of intervention i alarm group
  number of enuresis episodes (episodes per week)
change in Nocturia frequency | Change in number of nocturiaepisodes per night measured one week at Baseline (before intervention) and week 8 of intervention
  number of nocturia episodes/nights (nocturia episodes per night)

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Dept pediatrics, Aalborg University Hospital, Aalborg
  - dept Pediatrics, Aarhus University Hospital, Aarhus N
  - Børneafdelingen, Herning, Herning
  - Dept pediatrics, North Denmark Regional Hospital Hjoerring Hjoerring, Hjørring

IPD SHARING:
Plan to Share IPD: Undecided